CLINICAL TRIAL: NCT07365683
Title: A Prospective Randomized Non-blinded Study of Safety and Efficacy of Bilastine Up-dosing (40 mg) Versus Combination of Bilastine (20 mg) With Levocetrizine (5mg) in the Treatment of Chronic Spontaneous Urticaria
Brief Title: Efficacy of Bilastine Up-dosing (40 mg ) Versus Combination of Bilastine (20 mg )With Levocitirizine (5 mg) in the Treatment of Chronic Spontaneous Urticaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derma Techno Pakistan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IERC/DER/2024/01
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Spontaneous Urticaria (CSU)
Keywords: up-dosing +combination
MeSH Terms: conditions — Chronic Urticaria | interventions — bilastine; levocetirizine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (tab bilastine 40mg ) (Active Comparator): patients received oral tab bilastine 20 mg twice daily for 6 weeks
  Interventions: Drug: tab bilastine 20 mg
- Group B ( tab bilastine 20 mg + tab levocetrizine 5 mg ) (Active Comparator): patients received tab bilastine 20 mg in the morning and tab levocitrizine 5 mg in the evening for 6 weeks
  Interventions: Drug: tab bilastine 20 mg + tab levocetrizine 5 mg

INTERVENTIONS:
Drug: tab bilastine 20 mg — tab bilastine 20 mg given orally twice a day for 6 weeks
  Arms: Group A (tab bilastine 40mg )
Drug: tab bilastine 20 mg + tab levocetrizine 5 mg — tab levocitrizine 5 mg given orally at night with combination of tab bilastine 20 mg in the morning for 6 weeks
  Arms: Group B ( tab bilastine 20 mg + tab levocetrizine 5 mg )

SUMMARY:
This study aims to compare the effectiveness and safety of two commonly used antihistamines, bilastine 20 mg and levocetirizine 5 mg, in patients diagnosed with chronic urticaria. Chronic urticaria is a skin condition characterized by recurrent itchy wheals that significantly affect quality of life.

Eligible participants will be randomly assigned to receive either bilastine or levocetirizine for a defined treatment period. The severity of symptoms, improvement in itching and wheals, and any adverse effects will be assessed during follow-up visits.

The results of this study will help determine which treatment provides better symptom control with fewer side effects in patients with chronic urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of CSU as per operational definitions.
* Patients already taking Bilastine 20 mg and still getting new lesions.
* UAS7 score >3
* Age range of 18-70 years
* Both male and female patients

Exclusion Criteria:

* • women Patients who have already received treatment of CSU other than Bilastine.

  * Patients taking oral or topical corticosteroids
  * Pregnant or lactating
  * Patients with hereditary angioedema, atopic dermatitis, systemic immune disorders, collagen vascular diseases, immunocompromised status, Chronic liver or kidney failures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
change in urticaria severity score (UAS7) | baseline to 6 weeks
  change in urticaria severity score (UAS7) from baseline to 6 weeks UAS7 is a validated composite score assessing daily wheal number and pruritis severity over 7 consecutive days ,with total scores ranging from 0 to 42.
  Higher scores indicate more severe urticaria activity and a reduction in score reflects clinical improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- combined military hospital ,Okara, Okāra, Punjab Province, Pakistan